CLINICAL TRIAL: NCT03393637
Title: Mentors Offering Maternal Support (M-O-M-S™): A Prenatal Program Building Maternal Self-Esteem, Coping, and Resilience and Decreasing Depression.
Brief Title: Mentors Offering Maternal Support (M-O-M-S™): A Prenatal Program for Decreasing Maternal Anxiety and Depression
Acronym: M-O-M-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Incarnate Word (Other)
Collaborators: Joint Program Committee - 5 (Unknown); 59th Medical Wing (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency); Madigan Army Medical Center (U.S. Federal Agency); 711th Human Performance Wing (Unknown)
Responsible Party: Principal Investigator, Karen L. Weis, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWH20170069H
Record Dates: First submitted 2017-11-01; First posted 2018-01-08 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Anxiety Fear; Prenatal Depression; Infant, Low Birth Weight; Preterm Birth; Maternal
Keywords: prenatal anxiety; pregnancy; depression; military; intervention
MeSH Terms: conditions — Premature Birth; Depression

STUDY DESIGN:
Intervention Model Description: Following consent, the participants will randomized to either the treatment or control groups using a computer-generated randomization table developed prior to study start. They will be randomized to either the MOMS intervention or prenatal care without the MOMS. Women randomized to the MOMS program will be assigned to a MOMS group in the first trimester.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-O-M-S Intervention (Experimental): M-O-M-S intervention is 10, 1 hour prenatal mentored support groups
  Interventions: Behavioral: Mentors Offering Maternal Support (M-O-M-S)
- Routine Prenatal Care (No Intervention): Routine prenatal care in accordance with the Department of Defense Pregnancy Guidelines

INTERVENTIONS:
Behavioral: Mentors Offering Maternal Support (M-O-M-S) — 10, 1 hour, structured classes meeting every-other-week in person beginning in the first trimester of pregnancy and unlimited access to mentor support.
  Arms: M-O-M-S Intervention

SUMMARY:
The M-O-M-S project evaluates the effectiveness of the M-O-M-S program for improving birth outcomes and maternal-infant attachment and role satisfaction in a large military sample.

DETAILED DESCRIPTION:
The M-O-M-S project is a longitudinal, multi-site, randomized controlled trial to test program effectiveness for decreasing prenatal maternal anxiety and depression and increasing self-esteem and resilience and assess the relationship to pregnancy complications, birth outcomes, postpartum maternal-infant attachment, role satisfaction and parental stress.

ELIGIBILITY:
Inclusion Criteria:

* Prima or multigravida, first trimester of pregnancy at consent, greater than or equal to 18 years old, active duty, a wife of an active duty service member, or a retiree

Exclusion Criteria:

* Anticipated permanent change of station during the study (unless going to another one of the study sites or able to complete all treatment components prior to move), dependent daughter of active duty or retired military, greater than 12 weeks gestation at consent, less than 18 years of age and inability to understand English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant military women in the first trimester of pregnancy
Enrollment: 1717 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Lederman Self-Evaluation Questionnaire | assessing change between gestational weeks 12, 16, 24, and 32 of pregnancy
  Seven dimensions of pregnancy-specific anxiety
Rosenberg Self-Esteem Scale | assessing change between gestational weeks 12, 16, 24, and 32 of pregnancy and 1, 3, & 6 months postpartum
  10-item scale measuring the degree to which one values oneself
Family Adaptability and Cohesion Evaluation Scales | assessing change between gestational weeks 12, 16, 24, and 32 of pregnancy and 1, 3, & 6 months postpartum
  30-item instrument measuring the ability of the family (couple) to change its roles, rules, and power structure.
Edinburgh Postnatal Depression Scale | assessing change between gestational weeks 12, 16, 24, and 32 of pregnancy and 1, 3, & 6 months postpartum
  10-item scale measuring prenatal or postpartum symptoms of depression
Social Support Index | assessing change between gestational weeks 12, 16, 24, and 32 of pregnancy and 1, 3, & 6 months postpartum
  17-item scale measuring the extent to which families are integrated into the community, view the community as a source of support, and feel that the community can provide emotional, esteem, and network support
Family Index Coherence | assessing change between gestational weeks 12, 16, 24, and 32 of pregnancy and 1, 3, & 6 months postpartum
  17-item instrument measuring the degree to which families feel committed to the military mission and identify a subscale of family coping to manage life changes and stresses
Brief Resilience Scale | assessing change between gestational weeks 12, 16, 24, and 32 of pregnancy and 1, 3, & 6 months postpartum
  6-item instrument developed to measure the concept of "bouncing back from stress."
Postpartum Self-Evaluation Questionnaire | assessing change between 1, 3, & 6 months postpartum
  82-items measuring the woman's perceived postpartum adaptation to motherhood

SECONDARY OUTCOMES:
Infant birthweight | delivery weight of infant documented at delivery
  exact measure obtained from the delivery or infant record of the infants weight at birth in grams
Gestational age at birth | at first prenatal appointment up to 12 weeks
  Gestational age in weeks at birth determined from last menstrual period (LMP) and/or first trimester ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Weis, PhD, Principal Investigator — University of Kansas Medical Center
Locations (3):
- United States (3):
  - Naval Medical Center San Diego, San Diego, California
  - Joint Base San Antonio, San Antonio, Texas
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available to the local site PIs and to Department of Defense (DoD) OB Consultants. Study protocols are available upon request for DoD leaders within obstetrics.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be come available o/a February 2021
Access Criteria: As time approaches for complete data, will have available site with data.

REFERENCES:
- [Background] Weis KL, Ryan TW. Mentors offering maternal support: a support intervention for military mothers. J Obstet Gynecol Neonatal Nurs. 2012 Mar;41(2):303-314. doi: 10.1111/j.1552-6909.2012.01346.x. PMID 22834852
- [Background] Weis KL, Lederman RP, Lilly AE, Schaffer J. The relationship of military imposed marital separations on maternal acceptance of pregnancy. Res Nurs Health. 2008 Jun;31(3):196-207. doi: 10.1002/nur.20248. PMID 18213640
- [Result] Weis KL, Lederman RP, Walker KC, Chan W. Mentors Offering Maternal Support Reduces Prenatal, Pregnancy-Specific Anxiety in a Sample of Military Women. J Obstet Gynecol Neonatal Nurs. 2017 Sep-Oct;46(5):669-685. doi: 10.1016/j.jogn.2017.07.003. Epub 2017 Jul 24. PMID 28751158
- [Derived] O'Connell MA, Khashan AS, Leahy-Warren P, Stewart F, O'Neill SM. Interventions for fear of childbirth including tocophobia. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013321. doi: 10.1002/14651858.CD013321.pub2. PMID 34231203

DOCUMENTS (1):
  • Informed Consent Form (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT03393637/ICF_000.pdf